CLINICAL TRIAL: NCT02127281
Title: Randomized Controlled Trial of Wound Management With Negative Pressure Dressing Versus Standard Dressing After Knee and Hip Revision Arthroplasty.
Brief Title: Evaluation of Wound Management With Negative Pressure Dressing Versus Standard Dressing After Revision Arthroplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: KCI USA, Inc (Industry)
Responsible Party: Principal Investigator, Carlos Higuera-Rueda, Staff, Adult Reconstruction, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCF 14-273
Record Dates: First submitted 2014-04-29; First posted 2014-04-30 (Estimated); Results first posted 2018-03-26 (Actual); Last update posted 2018-09-19 (Actual); Status verified 2018-08

CONDITIONS: Prosthesis-related Infections; Wound Complications; Joint Diseases; Musculoskeletal Diseases
Keywords: Revision total knee arthroplasty; Revision total hip arthroplasty; Negative pressure wound therapy system (NPWT); Drainage
MeSH Terms: conditions — Prosthesis-Related Infections; Joint Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prevena (Active Comparator): Prevena NPWT system will be used immediately following surgery and continue postoperatively until hospital discharge (expected average of 4 days).
  Interventions: Device: Prevena
- Control (No Intervention): A standard of care sterile wound dressing will be placed.

INTERVENTIONS:
Device: Prevena — Device will be applied at end of procedure over closed incision.
  Arms: Prevena

SUMMARY:
The purpose of this study is to determine the efficacy of a negative pressure wound therapy (NPWT) system after revision total knee and hip arthroplasty in patients at high risk for infection. It is hypothesized that the use of NPWT system (i.e., Prevena) in high risk patients prevents wound complications and decreases reoperation rates.

DETAILED DESCRIPTION:
One of the primary causes of un-planned readmission following lower extremity arthroplasty procedures is infection. Continuous wound drainage poses a serious risk for infection and is often initially treated with absorbent dressings and/or oral antibiotics. Comorbidities such as obesity, diabetes and tobacco abuse predisposes to wound complications and therefore infection after these procedures. NPWT has proven to be effective for postoperative drainage and decreases the risk for infection or further reoperation. This prospective randomized trial will involve 160 patients at high risk for infection undergoing revision total knee or hip arthroplasty; 80 patients will be randomly selected to be treated with the NPWT system (Prevena) and randomly selected to be treated with the current standard of care wound dressing (control group). Patients will be enrolled at a single site of the Cleveland Clinic Health System (Main Campus).

ELIGIBILITY:
Inclusion Criteria:

* Scheduled revision Total Hip or Knee Arthroplasty Procedure
* Presence of one of the following: body mass index (BMI) greater than 35, use of blood thinners other than acetylsalicylic acid (ASA) after surgery, peripheral vascular disease, depression, diabetes mellitus, current tobacco use, history of prior infection, current use of immunomodulators or steroids, current history of cancer or hematological malignancy, rheumatoid arthritis, renal failure or dialysis, malnutrition, liver disease, transplant status, or HIV.

Exclusion Criteria:

* Patient lives >100 miles from hospital
* Patient is < 18 years old
* Silver allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-05; Primary Completion 2017-04-24 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Higuera-Rueda, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hansen E, Durinka JB, Costanzo JA, Austin MS, Deirmengian GK. Negative pressure wound therapy is associated with resolution of incisional drainage in most wounds after hip arthroplasty. Clin Orthop Relat Res. 2013 Oct;471(10):3230-6. doi: 10.1007/s11999-013-2937-3. PMID 23539123
- [Background] Bozic KJ, Kurtz SM, Lau E, Ong K, Chiu V, Vail TP, Rubash HE, Berry DJ. The epidemiology of revision total knee arthroplasty in the United States. Clin Orthop Relat Res. 2010 Jan;468(1):45-51. doi: 10.1007/s11999-009-0945-0. Epub 2009 Jun 25. PMID 19554385

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevena | Control
Started | 80 | 80
Completed | 79 | 80
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prevena | Control | Total
Number analyzed (Participants) | 80 | 80 | 160
Age, Continuous [Mean (Full Range); unit: years] | 65 [27 to 90] | 65 [37 to 93] | 65 [27 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 35 | 75
  Male | 40 | 45 | 85
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 65 | 66 | 131
  Non-white | 15 | 14 | 29
Body mass index [Mean (Full Range); unit: kg/m^2] | 31.9 [20.2 to 53.7] | 33.4 [20.4 to 58.7] | 32.7 [20.2 to 58.7]
Charlson comorbidity index [Count of Participants; unit: Participants] — The Charlson Comorbidity Index contains 19 categories of comorbidity and predicts the ten-year mortality for a patient who may have a range of co-morbid conditions. Each condition is assigned with a score of 1,2,3 or 6 depending on the risk of dying associated with this condition. A higher score indicated a higher level of illness.
  Participants
    0 | 32 | 24 | 56
    1 | 19 | 21 | 40
    >=2 | 29 | 35 | 64
American Society of Anesthesiologists score [Count of Participants; unit: Participants] — American Society of Anesthesiologists score a global score that assesses the physical status of patients before surgery, based on five classes 1 to 5. A higher score indicated a higher level of illness.
  Participants
    =<2 | 14 | 10 | 24
    >=3 | 66 | 70 | 136

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Wound Complications
Description: Any wound complications including but not limited to drainage, blisters, cellulitis, superficial infection, and deep infection.
Time Frame: Within 90 days after surgery
Population: 80 patients allocated to the prevena arm, and 79 patients were analyzed: 1 patient lost to follow-up; also, 1 patient had the prevena removed early but included as an intent to treat.
  80 patients allocated to control arm, with 80 patients analyzed. 6 patients did not receive the allocated treatment but were included for intent to treat
Measure: Number; unit: participants
Arm/Group | Prevena | Control
Number analyzed (Participants) | 79 | 80
participants | 9 | 22

2. Primary Outcome: Re-operation Rates
Description: Number of patients who required re-operations that were related to the revision arthroplasty and occurred within 90 days of the revision
Time Frame: Within 90 days after surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Control
Number analyzed (Participants) | 79 | 80
Participants | 5 | 11

3. Primary Outcome: Readmission Rates
Description: Number of patients who had hospital readmission(s) related to the revision surgery that occurred within 90 days of revision
Time Frame: Within 90 days after surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Control
Number analyzed (Participants) | 79 | 80
Participants | 16 | 16

4. Secondary Outcome: Knee Flexion
Description: Mean knee flexion (degrees) at 4 weeks postoperatively
Time Frame: 4 weeks postoperative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Prevena | Control
Number analyzed (Participants) | 27 | 31
degrees | 89.7 (21.6) | 88.9 (23.3)

5. Secondary Outcome: HOOS and KOOS Scores at 90 Days Postoperatively
Description: Mean Hip Osteoarthritis Outcome Score (HOOS), Knee Osteoarthritis Outcomes Score (KOOS) at 90 days postoperatively. Presented as subscores, including activities of daily living (ADL), pain, quality of life (QOL), symptoms, sports and recreation. All subscores range from 0-100, with 0 being the worst score and 100 being the best possible score.
Time Frame: 90 days postoperative
Population: The number analyzed is different from the overall number because there are separate questionnaires for Hip and Knee, and there were Hips and Knees in both the Prevena and Control groups
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prevena | Control
Number analyzed (Participants) | 79 | 80
units on a scale
  HOOS ADL: number analyzed (Participants) | 35 | 28
  HOOS ADL | 64.1 (23.9) | 66.4 (25.3)
  HOOS Pain: number analyzed (Participants) | 34 | 29
  HOOS Pain | 72.4 (23.7) | 70.3 (26.5)
  HOOS QOL: number analyzed (Participants) | 35 | 28
  HOOS QOL | 42.7 (21.3) | 37.9 (26.6)
  HOOS Symptoms: number analyzed (Participants) | 35 | 28
  HOOS Symptoms | 71.3 (17.4) | 70.2 (23.5)
  KOOS ADL: number analyzed (Participants) | 29 | 28
  KOOS ADL | 60.5 (24.7) | 54.3 (22.9)
  KOOS pain: number analyzed (Participants) | 29 | 29
  KOOS pain | 57.1 (24.9) | 55.8 (25.5)
  KOOS symptoms: number analyzed (Participants) | 29 | 27
  KOOS symptoms | 58.9 (18.1) | 55.9 (20.2)

6. Secondary Outcome: HOOS and KOOS Scores at 90 Days Postoperatively
Description: as for outcome 5
Time Frame: 90 days postoperative
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Prevena | Control
Number analyzed (Participants) | 79 | 80
units on a scale
  HOOS sports/rec: number analyzed (Participants) | 35 | 28
  HOOS sports/rec | 18.8 [6.3 to 34.4] | 21.9 [6.3 to 48.4]
  KOOS QOL: number analyzed (Participants) | 29 | 30
  KOOS QOL | 43.8 [25 to 62.5] | 34.4 [14.1 to 43.8]
  KOOS sports/rec: number analyzed (Participants) | 29 | 27
  KOOS sports/rec | 0 [0 to 25] | 10 [0 to 15]

7. Secondary Outcome: Timed-up-and-go Test
Description: Median Timed-up-and-go test (seconds)
Time Frame: 4 weeks postoperatively
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Prevena | Control
Number analyzed (Participants) | 53 | 39
seconds | 25 [14.3 to 37] | 24.2 [15 to 39.1]

8. Secondary Outcome: Hip Range of Motion (Flexion)
Description: Mean hip range of motion (flexion, in degrees) at 4 weeks postoperatively
Time Frame: 4 weeks postoperative
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Prevena | Control
Number analyzed (Participants) | 25 | 23
degrees | 73.6 (22.9) | 75.3 (25)

9. Secondary Outcome: VR-12 Questionnaire
Description: Mean VR-12 scores, presented as 2 composite scores physical component summary (PCS) and mental component summary (MCS). Physical Component Score (PCS): Provides greater emphasis on questions about general health, physical functioning and role playing and bodily pain. Mental Component Score (MCS): Provides greater emphasis on questions about role-emotional, vitality/mental health and social functioning. PCS and MCS summary scores are standardized using a z-score transformation and normed to a U.S. population (based on a 1990 norm) of a score of 50 and a standard deviation of 10. Higher MCS and PCS scores reflect better overall physical and mental health, respectively.
Time Frame: 90 days postoperatively
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Prevena | Control
Number analyzed (Participants) | 68 | 60
z-score
  PCS | 33.3 (9.6) | 31.5 (10.3)
  MCS | 50.2 (12.3) | 46.6 (14.1)

10. Secondary Outcome: Hip Range of Motion
Description: Median hip range of motion (extension, in degrees) at 4 weeks postoperatively
Time Frame: 4 weeks postoperative
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Prevena | Control
Number analyzed (Participants) | 24 | 22
degrees | 5 [0 to 10] | 0 [0 to 8]

11. Secondary Outcome: Knee Extension
Description: Median knee extension (degrees) at 4 weeks postoperatively
Time Frame: 4 weeks postoperative
Measure: Median (Inter-Quartile Range); unit: degrees
Arm/Group | Prevena | Control
Number analyzed (Participants) | 32 | 31
degrees | 5 [0 to 10] | 5 [0 to 10]

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Prevena | Control
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/80
Serious Adverse Events (participants affected / at risk) | 26/80 | 31/80
Other Adverse Events (participants affected / at risk) | 9/80 | 24/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevena (N=80) | Control (N=80)
Prosthetic Joint Infection (Infections and infestations) | 1 (1) | 2 (2)
Dislocation (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Venous Thrombosis (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Readmission (Investigations) | 16 (16) | 16 (16)
Reoperation (Investigations) | 5 (5) | 11 (11)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevena (N=80) | Control (N=80)
Wound drainage (Skin and subcutaneous tissue disorders) | 9 (9) | 22 (22)
mild edema (lung) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT02127281/Prot_SAP_000.pdf